CLINICAL TRIAL: NCT00614003
Title: Efficacy of a Training Intervention on the Quality of Case Coordinators and Nurses' Decision Support for Patients Deciding About the Place of Care at the End Of-Life: A Randomized Control Trial
Brief Title: Evaluation of an Intervention Designed to Enhance the Quality of Decision Support Provided to Patients Making Decisions About End-of-life Place of Care
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: H-01-07-09
Record Dates: First submitted 2008-01-18; First posted 2008-02-13 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Palliative Care
Keywords: decisional conflict;; decision quality;; place of end of life care;; provider education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): decision support
  Interventions: Behavioral: Decision support skills building Intervention

INTERVENTIONS:
Behavioral: Decision support skills building Intervention — Decision support skills

SUMMARY:
Most dying cancer patients would prefer a home death yet die in an institution. Patients can experience uncertainty when weighing practical considerations, concern for others, and their personal ratings about the desirability and undesirability of various outcomes related to different locations of care. Health professionals, trained in decision support, can help patients to make decisions that are informed by both relevant information and what outcomes are most valued by patients. Therefore, I will study if an educational intervention can help nurses and case managers to strengthen their skills and confidence in providing patient decision support around place of end of life care.

Project Description:

Using a two step approach I will study if the quality of providers decision support can be improved with an education. In step one nurses and care coordinators will be interviewed to identify factors that make it easier or more difficult to provide patient decision support. This information will be used to develop an education program. In step two, nurses and care coordinator volunteers will be assigned by a flip of a coin to either receive the decision support education or not. Before and after the education program the quality of the decision support participants provide will be measured and compared. As well, participants receiving the education program will be asked about their satisfaction with the education program.

DETAILED DESCRIPTION:
Most terminal cancer patients prefer home palliation yet die in an institution. Some experience decisional conflict when weighing options regarding place of care. Community Case Managers and Nurses are well positioned to identify decisional needs and provide decision support; however, they generally lack skills and confidence in doing so. This study aims to determine whether the quality of case managers' and nurses' decision support can be improved with a theory-based skills-building intervention.

In phase one a needs assessment will be conducted with about 20 key informants. In phase two, nurses will be randomly allocated to an intervention or control group. The intervention, informed by the needs assessment, is comprised of: an auto-tutorial; an interactive skills building workshop; a decision support protocol; performance feedback, and educational outreach.

Participants will be assessed: a) at baseline (quality of decision support); b) after the auto-tutorial (knowledge); and six to eight weeks after the other interventions (quality of decision support; confidence and intention to integrate decision support into practice). Between group differences in the primary outcome (quality of decision support scores) will be analyzed using a repeated measures ANOVA.

ELIGIBILITY:
Inclusion Criteria:

Nurses and case coordinators who:

* are members of a regulated health profession
* care for palliative cancer patients, and/or
* cancer patients with advanced disease, and
* work at least 4 shifts per month,
* in a clinical area where end of life care discussions are likely to be undertaken, and
* are proficient in written and spoken English.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2007-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Decision support quality audit using simulated patients measured by the validated and reliable Decision Support Analysis Tool | 6 month

SECONDARY OUTCOMES:
Knowledge of place of care determinants and decision support concepts; self perceived quality of decision support provision in clinical practice and behavior intention survey; acceptability and utility of intervention components | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Annette O'Connor, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (5):
- Canada (5):
  - St. Elizabeths Health Care Agency, Kingston, Ontario
  - Ottawa Carefor Nursing Services, Ottawa, Ontario
  - SCOHS Regional Palliative Care Community Services, Ottawa, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Community Care Access Center's (CCAC), Toronto, Ontario

REFERENCES:
- [Derived] Murray MA, O'Connor A, Stacey D, Wilson KG. Efficacy of a training intervention on the quality of practitioners' decision support for patients deciding about place of care at the end of life: A randomized control trial: Study protocol. BMC Palliat Care. 2008 Apr 30;7:4. doi: 10.1186/1472-684X-7-4. PMID 18447916